CLINICAL TRIAL: NCT04688021
Title: A Single-arm, Single-center Trial of Prophylactic Tocilizumab for Acute GVHD Prevention After Haploidentical HSCT.
Brief Title: A Single-arm Trial of Prophylactic Tocilizumab for Acute GVHD Prevention After Haploidentical HSCT.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yi Luo (Other)
Responsible Party: Sponsor-Investigator, Yi Luo, Clinical Professor, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TZ-001
Record Dates: First submitted 2020-12-11; First posted 2020-12-29 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Leukemia; Graft-versus-host-disease
Keywords: hematopoietic stem cell transplantation; graft-versus-host disease
MeSH Terms: conditions — Leukemia; Graft vs Host Disease | interventions — Cytarabine; Busulfan; Cyclophosphamide; Semustine; thymoglobulin; tocilizumab; Cyclosporine; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocilizumab cohort (Experimental): Each patient receives Tocilizumab (8 mg/kg, i.v.) on day -1 added to conventional acute GVHD prophylaxis regimen (CsA+MTX+low-dose MMF+ATG) of haploidentical HSCT.
  Interventions: Drug: Cytarabine; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Me-CCNU; Drug: Rabbit antithymocyte globulin; Drug: Tocilizumab; Procedure: Allogeneic HSCT; Drug: Cyclosporin A; Drug: Mycophenolate Mofetil; Drug: MTX

INTERVENTIONS:
Drug: Cytarabine — 4 mg/m2/day administered IV day -10 through -9.
Drug: Busulfan — 3.2 mg/kg/day administered IV day -8 through -6.
Drug: Cyclophosphamide — 1.8 g/m2/day administered IV day -5 through -4.
Drug: Me-CCNU — 250mg/m2 once administered orally on day -3.
Drug: Rabbit antithymocyte globulin — 1.5mg/kg/day administered IV day -5 through -2.
Drug: Tocilizumab — 8mg/kg administered IV on day -1.
Procedure: Allogeneic HSCT — Day 0
Drug: Cyclosporin A — 2.5 mg/kg/day administered intravenously from day -7, target: 200-300ng/mL. Usually tapered during the second month, and ended in complete withdrawal during the ninth month after transplantation.
Drug: Mycophenolate Mofetil — 500 mg/day administered intravenously from day -9, ended in complete withdrawal on day +100.
Drug: MTX — 15 mg/m2 administered intravenously on day +1, 10mg/m2 on day +3, +6, and +9.

SUMMARY:
A single-arm trial using Tocilizumab for acute GVHD prophylaxis after haploidentical HSCT.

DETAILED DESCRIPTION:
This study will enroll haploidentical HSCT patients with high risk for acute GVHD. Tocilizumab (8mg/kg) will be added to the conventional acute GVHD prophylaxis regime (CsA+Methotrexate(MTX)+low dose mycophenolate mofetil(MMF)+ATG) on day -1 of transplant. The previous patients will be used as control.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematological malignancies in complete remission (CR) who are eligible and planned for haploidentical HSCT. The donor specific antibody is negative
* Patient age 16-60 years
* Mother donor, or female donor (age >50) for female-male transplant
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Creatinine clearance rate > 60 mL/min (estimate by Cockcroft-Gault Equation)
* alanine transaminase (ALT) and aspartate aminotransferase (AST)≤ 2.5×upper limit of normal (ULN), and total bilirubin ≤ 1.5×ULN （upper limit of normal, ULN）
* Left ventricular ejection fraction (LVEF) ≥50% as measured by echocardiography
* Acceptation to sign the informed consent

Exclusion Criteria:

* History of previous HSCT
* Present active infection (including bacterial, virus or fungal)
* History of Tocilizumab infection
* History of inflammatory bowel disease
* History of demyelinating disease
* Patients who are HIV-positive, or with uncontrolled chronic hepatitis B virus (HBsAg positive) or hepatitis C virus (anti-HCV) infections
* Women who are pregnant (β-chorionic gonadotropin+) or breast feeding
* Refusal to sign the informed consent

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2024-12-03 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of grade II-IV acute graft-versus-host disease | 100 days
  Date of symptom onset, maximum clinical grade, and dates and types of treatment will be recorded. Dates of symptom onset of grade II-IV acute graft-versus-host disease (aGVHD) will be recorded. The aGVHD score of each affected organ will be recorded.
Cumulative incidence of non grade II-IV acute graft-versus-host disease survival | 100 days
  All patients will be tracked from Day 0 to date of grade II-IV acute graft-versus-host disease (aGVHD) onset. Patients who did not present grade II-IV aGVHD or died will be censored at the last date they were assessed and deemed free of grade II-IV aGVHD.

SECONDARY OUTCOMES:
Cumulative incidence of engraftment | 100 days
  All patients will be tracked from Day 0 to date of myeloid and platelet engraftments, respectively.
Cumulative incidence of infections | 2 years
  All patients will be tracked from Day 0 to date of infection diagnosis as proved by relevant standard diagnostic criteria.
Overall survival (OS) | 2 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Progression-free survival (PFS) | 2 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Cumulative incidence of transplant-related nonrelapse mortality (NRM) | 2 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.
Cumulative incidence of disease relapse or progression | 2 years
  All patients will be tracked from Day 0 to date of first objective disease progression, death from any cause, or last patient evaluation. Patients who have not progressed or died will be censored at the last date they were assessed and deemed free of relapse or progression.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No